CLINICAL TRIAL: NCT01920737
Title: A Novel "Pediatric-Inspired" Regimen With Reduced Myelosuppressive Drugs for Adults (Aged 18-60) With Newly Diagnosed Ph Negative Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Shire (Industry); Duke University (Other); Weill Medical College of Cornell University (Other); Lehigh Valley Health Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-266
Record Dates: First submitted 2013-08-07; First posted 2013-08-12 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Leukemia
Keywords: ALL; Bone Marrow; Ph Negative; Daunorubicin; Vincristine; Prednisone; PEG-Asparaginase; Methotrexate; 16-MP (6-Mercaptopurine); Cyclophosphamide; Cytarabine; Leucovorin; Dexamethasone; 12-266
MeSH Terms: conditions — Leukemia | interventions — Daunorubicin; Vincristine; Prednisone; pegaspargase; Methotrexate; Mercaptopurine; Cyclophosphamide; Cytarabine; Leucovorin; Dexamethasone; Blood Specimen Collection; Positron Emission Tomography Computed Tomography

ARMS (1):
- Leukemia Patients (Experimental): The treatment plan has 6 treatment cycles. The cycle names are listed in the following order:
  Induction Phase I - Induction Phase II - Intensification I - Re-induction I - Intensification II - Re-induction II Each cycle is given over a period of 4-6 weeks and the interval between them can range between 1-3 weeks. Based the patients medical condition, the doctor may decide to change the timing of the drugs, the interval between the drugs in a cycle, or the interval between the cycles. After receiving all cycles you will continue with a 36 months treatment part that is called Maintenance.
  Interventions: Drug: Daunorubicin; Drug: Vincristine; Drug: Prednisone; Drug: PEG-Asparaginase; Drug: Methotrexate; Drug: 6-MP (6-Mercaptopurine); Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Leucovorin; Drug: Dexamethasone; Other: Blood draw; Device: CT/PET scans

INTERVENTIONS:
Drug: Daunorubicin — In the event of a shortage of daunorubicin, doxorubicin may be used as a substitute.
Drug: Vincristine
Drug: Prednisone
Drug: PEG-Asparaginase
Drug: Methotrexate
Drug: 6-MP (6-Mercaptopurine)
Drug: Cyclophosphamide
Drug: Cytarabine
Drug: Leucovorin
Drug: Dexamethasone
Other: Blood draw
Device: CT/PET scans — PET or CT scan every 6 months for 3 years

SUMMARY:
The purpose of the study is to find out whether the combination of chemotherapy drugs that are routinely used in children with ALL, will be safe and effective in treating adult patients with ALL. The standard treatment for adults with ALL consists of many chemotherapy drugs that are given in different combinations and in several steps. In adult ALL there is no standard which drugs to give and how to combine them. Some leukemias have a chromosome abnormality called Philadelphia chromosome (also called Ph Positive) and some leukemias do not (called Ph Negative). In this study we want to see whether this combination of chemotherapy drugs will be safe and effective in treating adult patients with Ph Negative ALL.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated Ph negative precursor B-cell or T-cell ALL confirmed by conventional flow cytometry or immunohistochemical stain Patients who have untreated B-cell or T-cell ALL confirmed by conventional flow cytometry or immunohistochemical stain, but Ph status is unknown, may also enroll.
* Patients with T-cell or B cell lymphoblastic lymphoma confirmed by conventional immature T- or pre B cell markers even if the bone marrow is not involved are also eligible
* Age 18 - 60 years
* ECOG performance status of 0-2
* Adequate renal function as demonstrated by a serum creatinine ≤ 2.0 mg/dl or a creatinine clearance of > 60 ml/min.
* Adequate hepatic function as demonstrated by a total bilirubin < 2.0 mg/dl (unless attributable to Gilbert's disease) and an alkaline phosphatase, AST, and ALT ≤ 4 times the upper limit of normal (unless clinically considered to be related to liver involvement with leukemia
* Normal cardiac function as demonstrated by a left ventricular ejection fraction ≥ 50% on echocardiogram or MUGA scan
* Negative serum pregnancy test in women of childbearing potential
* Men and women of childbearing potential must be willing to practice an effective method of birth control during treatment and at least 4 months after treatment is finished.
* Patients with central nervous system involvement by ALL are eligible and may receive concomitant treatment with radiation therapy and/or intrathecal chemotherapy in accordance with standard medical practice. For patients with CNS disease, dexamethasone may be temporarily administered instead of prednisone to reduce CNS pressure, at the discretion of the treating physician and after discussion with the MSK PI. Once dexamethasone is no longer needed, prednisone should be given as per protocol for 28 days.

Exclusion Criteria:

* Previous treatment for ALL, except for prior steroids and/or hydroxyurea
* Patients known to have Philadelphia (Ph)+ ALL are not eligible. Leukemia cell samples will be obtained from all patients enrolled before starting protocol treatment and submitted for Philadelphia chromosome testing by either karyotyping, or for bcr/abl1 translocation by FISH or by PCR for bcr/abl1. Patients who are later found to have Ph+ ALL should have treatment on this trial discontinued and will not be considered in the evaluation
* Lymphoid blastic crisis of chronic myelogenous leukemia
* Mature B-cell (Burkitt's) ALL
* Active serious infections not controlled by antibiotics
* Pregnant women or women who are breast-feeding
* Concurrent active malignancy requiring immediate therapy
* Clinically significant cardiac disease (NY Heart Association Class III or IV), including chronic arrhythmias, or pulmonary disease
* Known HIV positive status
* Other serious or life-threatening conditions deemed unacceptable by the principal investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-08-07; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
rate of molecular remission | 1 year
  i.e. minimal residual disease (MRD) negative status, as assessed by PCR and flow cytometry in the bone marrow after phase I induction.

SECONDARY OUTCOMES:
complete remission (CR) | 1 year
  All three criteria must be met for clinical complete remission:
  * Peripheral Blood Counts. The absolute neutrophil count should be ≥1,000/μl (sustained without growth factor support), and platelet count should be ≥100,000/μl (without transfusions), and no circulating blasts. After Induction remission assessment, blood counts are considered recovered at ANC ≥ 1,000 and PLT ≥75,000.
  * Bone Marrow Aspirate. Bone marrow cellularity should be approximate normal with evidence of maturation of all cell lineages and should contain <5% blasts.
  * Extramedullary Leukemia, such as CNS or soft tissue involvement, must not be present. If the patient had CNS involvement by ALL at the time of starting the study, the CNS involvement should be re-examined and interval determined by the treating physicians in order to determine if clinical complete remission
overall survival (OS) | 1 year
  OS will be calculated from the start of induction therapy to death or last follow-up.
event-free survival (EFS) | 1 year
  EFS survival will be calculated from the start of induction therapy to relapse (molecular or clinical), death, or last follow-up.
disease free survival (DFS) rates | 1 year
  DFS will be calculated from the time of clinical CR (or better) to relapse (molecular or clinical), death, or last follow-up.
minimal residual disease (MRD) status | 1 year
  Molecular relapse is defined as the conversion of RT-PCR from MRD negative to MRD positive on two consecutive tests performed on bone marrow at least one week apart, while still meeting criteria for clinical CR.
safety | 1 year
  Number of participants with adverse events. Frequencies of toxicities based on the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Geyer MB, Ritchie EK, Rao AV, Vemuri S, Flynn J, Hsu M, Devlin SM, Roshal M, Gao Q, Shukla M, Salcedo JM, Maslak P, Tallman MS, Douer D, Park JH. Pediatric-inspired chemotherapy incorporating pegaspargase is safe and results in high rates of minimal residual disease negativity in adults up to age 60 with Philadelphia chromosome-negative acute lymphoblastic leukemia. Haematologica. 2021 Aug 1;106(8):2086-2094. doi: 10.3324/haematol.2020.251686. PMID 33054114
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/